CLINICAL TRIAL: NCT03172416
Title: Phase 1 Study of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) With Oxaliplatin. Phase 1 Study of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) With Oxaliplatin and in Combination With Nivolumab in Patients With Peritoneal Carcinomatosis (PIANO)
Brief Title: Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) With Oxaliplatin In Patients With Peritoneal Carcinomatosis
Acronym: PIPAC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB 2016/01088
Record Dates: First submitted 2017-01-23; First posted 2017-06-01 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Peritoneal Carcinomatosis
Keywords: Gastric Cancer; Unresectable Peritoneal Carcinomatosis; Oxaliplatin; Pressurized intraperitoneal aerosol chemotherapy; Nivolumab
MeSH Terms: conditions — Peritoneal Neoplasms; Stomach Neoplasms | interventions — Oxaliplatin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oxaliplatin (Other): 3+3 dose escalation of oxaliplatin
  This is a single arm phase I trial in a 3 + 3 dose escalation and cohort expansion design evaluating the safety and tolerability of PIPAC using oxaliplatin.
  The pre-planned dose levels of oxaliplatin are 45mg/m2 (Cohort 1), 60mg/m2 (Cohort 2), 90mg/m2 (Cohort 3),120mg/m2 (Cohort 4) and 150mg/m2 (Cohort 5) administered as PIPAC. Successive cohorts of patients (3 participants/cohort) will be enrolled and started on a fixed dose of oxaliplatin. The protocol specifies oxaliplatin 45mg/m2 once every 6 weeks for Cohort 1. Dose escalation continues until dose-limiting toxicities (DLT) are observed in one-third of participants. If no DLT occurs, the next cohort will be enrolled at the next planned dose level. If 1 DLT occurs in a cohort, another 3 patients will be treated with the same dose level.
  Oxaliplatin every 6 weeks with IV nivolumab every 2 weeks
  PIPAC oxaliplatin at 90mg/m2 every 6 weeks with IV nivolumab at 240mg every 2 weeks
  Interventions: Drug: Oxaliplatin; Drug: Oxaliplatin & Nivolumab

INTERVENTIONS:
Drug: Oxaliplatin — This study started as a prospective, single arm phase I trial in a 3 + 3 dose escalation evaluating the safety and tolerability of PIPAC using oxaliplatin in patients with peritoneal carcinomatosis.
Drug: Oxaliplatin & Nivolumab — PIPAC oxaliplatin 90mg/m2 has been well tolerated in our Cohort 1 study. Hence, we added a second cohort (Cohort 2) which combines PIPAC oxaliplatin at 90mg/m2 every 6 weeks with IV nivolumab at 240mg every 2 weeks to evaluate the safety and tolerability of combination therapy.

SUMMARY:
PIPAC is a procedure that involves the administration of intraperitoneal chemotherapy using an innovative concept that enhances the efficacy by taking advantage of the physical properties of gas and pressure. The chemotherapy drugs will be delivered in aerosolised form. This results in a superior distribution and depth of penetration of the drug.

This research study serves to determine the safety profile and tolerability of PIPAC with oxaliplatin. It may offer a novel and effective option of treatment for patients with peritoneal carcinomatosis, who, at present have limited options involving the use of systemic chemotherapy and who suffer from poor life expectancy and poor quality of life.

To date, most trials have used PIPAC cisplatin with doxorubicin, or oxaliplatin alone, and more studies are on-going globally.

Intravenous (IV) nivolumab has been approved for the treatment of progressive gastric cancer after conventional chemotherapy. PIPAC in combination with nivolumab may have the potential to improve immune activation and response to immune checkpoint inhibition for patients with peritoneal disease.

Hence we propose an amendment to our trial protocol for the addition of a second cohort (Cohort 2) to investigate the safety and tolerability of the combination of PIPAC oxaliplatin and IV nivolumab.

DETAILED DESCRIPTION:
Gastric cancer is the 5th most common cancer (1 million incidences per year) and the third leading cause of cancer-related mortality worldwide (740,000 deaths per year). Unresectable gastric cancer is associated with a poor 5-year survival rate (< 30%) because of its late presentation with approximately 50% of the patients diagnosed at advanced stage with a median survival of about 12 months. The treatment for advanced gastric cancer patients relies mainly on doublet or triplet chemotherapy, but results are often limited by severe side effects of the aggressive regimens. Novel efficacious treatments with reduced adverse effects are highly desirable to improve the clinical outcome.

Peritoneal disease is notoriously difficult to treat. In patients with histologically proven unresectable or recurrent gastric cancer limited to the peritoneum and/or cancer cells in peritoneal cytology, the combination of intraperitoneal (IP) paclitaxel with systemic chemotherapy seems promising. However, a phase III trial (PHOENIX-GC trial) comparing IP regimen with systemic chemotherapy versus systemic therapy alone in Japan did not show any superiority of the IP regimen.

PIPAC is an innovative intraperitoneal chemotherapy concept that enhances the efficacy by taking advantage of the physical properties of gas and pressure. This results in a superior distribution and depth of penetration of the drug. A recent systematic review of 45 clinical studies on 1810 PIPAC procedures showed response rates of 50-91% for gastric cancer (median survival of 8 to 15 months), 71-86% for colorectal cancer (median survival of 16 months).

To date, most phase II trials utilising PIPAC involve the use of cisplatin and doxorubicin or oxaliplatin. Oxaliplatin is an approved drug for systemic chemotherapy, with well documented use intraperitoneally via hyperthermic intraperitoneal chemotherapy (HIPEC) as well. This makes is a favourable agent for PIPAC in early phase studies. The dose of oxaliplatin utilised for PIPAC in the literature has thus far been arbitrarily set at 92 mg/m2, which is approximately 80% of the drug concentration used in HIPEC. Furthermore, these studies were performed on patients with a recent or concurrent administration of systemic chemotherapy, which may make interpretation of the side effects and safety profile difficult to interpret.

In Cohort 1 of this study, we intend to determine the safety profile and tolerability of PIPAC with oxaliplatin by assessment of dose limiting toxicities and the adverse event profile.

Cancer immunotherapy with checkpoint inhibitor has demonstrated clinical activities and survival benefits as a monotherapy and in combination with other immunotherapies or conventional chemotherapies in multiple cancer types. Nivolumab has been showed to have overall survival benefit over placebo in the third line treatment of metastatic gastric cancer with a response rate of 11%. In the CheckMate032 trial, nivolumab, with or without ipilumumab, demonstrated durable responses and long-term survival. Nivolumab alone, dosed at 3mg/kg, had a response rate of 12%.

It is hypothesized that the delivery of PIPAC deep into the peritoneal tissue is likely to affect the tumor microenvironment and potentially release neoantigens which would improve clinical outcomes with immune checkpoint inhibition. Hence we propose an amendment to our trial protocol for the addition of a second cohort (Cohort 2) to combine this Phase I proof-of-concept study with nivolumab.

The aim is to determine the determine the safety profile and tolerability of PIPAC oxaliplatin by assessment of dose limiting toxicities and the adverse event profile. With Cohort 2, the co-primary endpoints are the safety and efficacy of the combination of PIPAC oxaliplatin and IV nivolumab. Safety will be evaluated in terms of adverse events, serious adverse events, discontinuation of treatment due to toxicity. Efficacy will be evaluated in terms of the percentage of patients with 6 months of time-to-treatment failure (TTF). TTF is defined as the interval from treatment initiation to treatment discontinuation for disease progression, treatment toxicity, and death. The secondary objective is to evaluate the clinical and pathological response of PIPAC oxaliplatin as well as to identify the pharmacokinetic profile of oxaliplatin administered via PIPAC. The clinical and pathological response to combination treatment will also be determined. Quality of life will be evaluated.

ELIGIBILITY:
Inclusion Criteria for Cohort 1:

* Gastric cancer patients with peritoneal metastasis on peritoneal cytology/histology.
* Patients who refuse, are unable to tolerate, or have completed at least 1st line systemic chemotherapy.
* Patients who have completed chemotherapy/targeted therapy > 21 days or at least 5 half-lives (or whichever is longer) prior to PIPAC.
* Age >21 years.
* Eastern Cooperative Oncology Group performance status 0-1.
* Adequate bone marrow function (neutrophil count >1500/mm3, hemoglobin >8.0 g/dl and platelet count >100 000/mm3).
* Adequate liver function (bilirubin, AST/ALT within upper limit of normal)
* Adequate renal function (serum creatinine within the upper limit of normal)
* Expected survival >3 months
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria for Cohort 1:

* Predominant extra-peritoneal metastases at the discretion of the study team after discussion at the multidisciplinary tumour board
* Good response to systemic chemotherapy based on RECIST guidelines VI.I with complete or partial response to systemic chemotherapy.
* Known allergy to oxaliplatin
* Previous malignancy unrelated to current peritoneal carcinomatosis diagnosed in the last 5 years
* Patients with treated skin cancer besides melanoma may be included.
* Patients with reproductive potential who refuse to use an adequate means of contraception (including male patients)
* Significant disease or conditions which, in the investigator's opinion, would exclude patient from the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating female

Inclusion Criteria for Cohort 2:

* Gastric cancer patients with peritoneal metastasis on peritoneal cytology/histology, for whom oxaliplatin is considered standard of care for the peritoneal carcinoma of origin.
* Patients who refuse, are unable to tolerate, or have completed at least 1st line systemic chemotherapy
* Patients who have completed chemotherapy/targeted therapy > 21 days or at least 5 half-lives (or whichever is longer) prior to PIPAC
* Patients must have recovered (≤ grade 1) from all reversible treatment toxicity from prior chemotherapy, radiotherapy or surgery.
* Age ≥21 years
* Eastern Cooperative Oncology Group performance status 0-1
* Adequate bone marrow function (neutrophil count ≥1500/mm3, hemoglobin ≥8.0 g/dl and platelet count ≥100 000/mm3)
* Adequate liver function (bilirubin ≤ 1.5x ULN(upper limit normal) and AST/ALT ≤3x ULN or ≤5x ULN in the presence of liver metastases)
* Adequate renal function (serum creatinine ≤1.5x ULN)
* Expected survival >3 months
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria for Cohort 2:

* Predominant extra-peritoneal metastases at the discretion of the study team after discussion at the multidisciplinary tumour board
* Patients who have previously received prior nivolumab or PD-/L1 blockade therapy
* Patients with clinical or radiological evidence of hollow viscera perforation or impending perforation, including but not limited to gastric, small bowel, colon, gallbladder. Decision will be made at the discretion of the study team in consultation with multidisciplinary tumour board or with necessary specialists
* Good response to systemic chemotherapy based on RECIST guidelines VI.I with complete or partial response to systemic chemotherapy.
* Active autoimmune disease requiring disease-modifying therapy.
* Concurrent systemic steroid therapy higher than physiologic dose (equivalent of prednisolone 10mg daily), except for short courses (< 2 weeks) required to treat acute medical conditions (e.g. asthma exacerbation, or for CT scans)
* Any form of active primary or secondary immunodeficiency.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled hypertension (systolic >160 mmHg and/or diastolic >100 mmHg), symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction/cerebrovascular event (≤ 6 months prior to study entry), cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, long term systemic immunosuppressant or corticosteroid, and active viral hepatitis.
* Known allergy to oxaliplatin
* Previous malignancy unrelated to current peritoneal carcinomatosis diagnosed in the last 2 years
* Patients with treated skin cancer besides melanoma may be included.
* Patients with reproductive potential who refuse to use an adequate means of contraception (including male patients)
* Significant disease or conditions which, in the investigator's opinion, would exclude patient from the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating female

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2017-04-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety Profile of PIPAC with oxaliplatin by monitoring adverse event profile of patient undergo PIPAC | 1 to 2 years
Tolerability of PIPAC with oxaliplatin by monitoring dose limiting toxicities | 1-2 years
Safety Profile of PIPAC with oxaliplatin in combination with IV nivolumab by monitoring adverse event profile of patient undergo PIPAC | 1-2 years
Tolerability of PIPAC with oxaliplatin in combination with IV nivolumab by monitoring dose limiting toxicities | 1-2 years

SECONDARY OUTCOMES:
Clinical response of PIPAC with oxaliplatin according to Peritoneal Cancer Index (PCI) | 1-2 years
Pathological response of PIPAC with oxaliplatin according to Peritoneal Regression Grade Scoring (PRGS) System | 1-2 years
Maximum concentration (Cmax) of oxaliplatin administered via PIPAC using blood drawn from patient. | Pre-dose; 30 and 45 minutes; and 1, 2, 4, 8, 24 and 30 hours
  Maximum concentration (Cmax) of oxaliplatin, for patients with peritoneal carcinomatosis after PIPAC administration.
Half-life (t1/2) of oxaliplatin administered via PIPAC using blood drawn from patient. | Pre-dose; 30 and 45 minutes; and 1, 2, 4, 8, 24 and 30 hours
  Half-life (t1/2) of oxaliplatin for patients with peritoneal carcinomatosis after PIPAC administration.
Area under the curve (AUC) of oxaliplatin administered via PIPAC using blood drawn from patient. | Pre-dose; 30 and 45 minutes; and 1, 2, 4, 8, 24 and 30 hours
  Area under the curve (AUC) of oxaliplatin for patients with peritoneal carcinomatosis after PIPAC administration
Clinical response of PIPAC with oxaliplatin in combination with IV nivolumab according to Peritoneal Cancer Index (PCI) | 1-2 years
Pathological response of PIPAC with oxaliplatin in combination with IV nivolumab according to Peritoneal Regression Grade Scoring (PRGS) System | 1-2 years
Maximum concentration (Cmax) of oxaliplatin and in combination with IV nivolumab administered via PIPAC using blood drawn from patient. | Pre-dose, 30 minutes, 1 and 30 hours
  Maximum concentration (Cmax) of oxaliplatin and in combination with IV nivolumab for patients with peritoneal carcinomatosis after PIPAC administration.
Half-life (t1/2) of oxaliplatin and in combination with IV nivolumab administered via PIPAC using blood drawn from patient. | Pre-dose, 30 minutes, 1 and 30 hours
  Half-life (t1/2) of oxaliplatin and in combination with IV nivolumab for patients with peritoneal carcinomatosis after PIPAC administration.
Area under the curve (AUC) of oxaliplatin and in combination with IV nivolumab administered via PIPAC using blood drawn from patient. | Pre-dose, 30 minutes, 1 and 30 hours
  Area under the curve (AUC) of oxaliplatin and in combination with IV nivolumab for patients with peritoneal carcinomatosis after PIPAC administration

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy So, MBChB, Principal Investigator — National University Hospital, Singapore
Locations (3):
- Ghent University Hospital, Ghent, Belgium
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishigami H, Kitayama J, Kaisaki S, Hidemura A, Kato M, Otani K, Kamei T, Soma D, Miyato H, Yamashita H, Nagawa H. Phase II study of weekly intravenous and intraperitoneal paclitaxel combined with S-1 for advanced gastric cancer with peritoneal metastasis. Ann Oncol. 2010 Jan;21(1):67-70. doi: 10.1093/annonc/mdp260. Epub 2009 Jul 15. PMID 19605503
- [Background] Solass W, Hetzel A, Nadiradze G, Sagynaliev E, Reymond MA. Description of a novel approach for intraperitoneal drug delivery and the related device. Surg Endosc. 2012 Jul;26(7):1849-55. doi: 10.1007/s00464-012-2148-0. Epub 2012 May 12. PMID 22580869
- [Background] Solass W, Herbette A, Schwarz T, Hetzel A, Sun JS, Dutreix M, Reymond MA. Therapeutic approach of human peritoneal carcinomatosis with Dbait in combination with capnoperitoneum: proof of concept. Surg Endosc. 2012 Mar;26(3):847-52. doi: 10.1007/s00464-011-1964-y. Epub 2011 Nov 1. PMID 22042585
- [Background] Robella M, Vaira M, De Simone M. Safety and feasibility of pressurized intraperitoneal aerosol chemotherapy (PIPAC) associated with systemic chemotherapy: an innovative approach to treat peritoneal carcinomatosis. World J Surg Oncol. 2016 Apr 29;14:128. doi: 10.1186/s12957-016-0892-7. PMID 27125996
- [Background] Solass W, Kerb R, Murdter T, Giger-Pabst U, Strumberg D, Tempfer C, Zieren J, Schwab M, Reymond MA. Intraperitoneal chemotherapy of peritoneal carcinomatosis using pressurized aerosol as an alternative to liquid solution: first evidence for efficacy. Ann Surg Oncol. 2014 Feb;21(2):553-9. doi: 10.1245/s10434-013-3213-1. Epub 2013 Sep 5. PMID 24006094
- [Background] Demtroder C, Solass W, Zieren J, Strumberg D, Giger-Pabst U, Reymond MA. Pressurized intraperitoneal aerosol chemotherapy with oxaliplatin in colorectal peritoneal metastasis. Colorectal Dis. 2016 Apr;18(4):364-71. doi: 10.1111/codi.13130. PMID 26400556
- [Derived] Sundar R, Chia DKA, Zhao JJ, Lee ARYB, Kim G, Tan HL, Pang A, Shabbir A, Willaert W, Ma H, Huang KK, Hagihara T, Tan ALK, Ong CJ, Wong JSM, Seo CJ, Walsh R, Chan G, Cheo SW, Soh CCC, Callebout E, Geboes K, Ng MCH, Lum JHY, Leow WQ, Selvarajan S, Hoorens A, Ang WH, Pang H, Tan P, Yong WP, Chia CSL, Ceelen W, So JBY. Phase I PIANO trial-PIPAC-oxaliplatin and systemic nivolumab combination for gastric cancer peritoneal metastases: clinical and translational outcomes. ESMO Open. 2024 Sep;9(9):103681. doi: 10.1016/j.esmoop.2024.103681. Epub 2024 Sep 16. PMID 39288528
- [Derived] Kim G, Tan HL, Chen E, Teo SC, Jang CJM, Ho J, Ang Y, Ngoi NYL, Chee CE, Lieske B, Shabbir A, Wang LZ, So JBY, Yong WP. Study protocol: phase 1 dose escalating study of Pressurized Intra-Peritoneal Aerosol Chemotherapy (PIPAC) with oxaliplatin in peritoneal metastasis. Pleura Peritoneum. 2018 Aug 29;3(3):20180118. doi: 10.1515/pp-2018-0118. eCollection 2018 Sep 1. PMID 30911663